CLINICAL TRIAL: NCT00594568
Title: Effect of γ-Secretase Inhibition on the Progression of Alzheimer's Disease: LY450139 Versus Placebo
Brief Title: Effect of LY450139 on the Long Term Progression of Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7666; H6L-MC-LFAN (Other: Eli Lilly and Company); CTRI/2009/091/000090 (Registry Identifier: India)
Record Dates: First submitted 2008-01-11; First posted 2008-01-15 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — N2-((2S)-2-(3,5-difluorophenyl)-2-hydroxyethanoyl)-N1-((7S)-5-methyl-6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-L-alaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo orally once daily for the first 76 weeks. At the end of 76 weeks, placebo arm participants received LY450139 titrated up to 140 milligrams (mg) orally once daily until Week 88.
  Interventions: Drug: Placebo
- 100 mg LY450139 (Experimental): Participants received 60 mg LY450139 orally once daily for 2 weeks, followed by 100 mg LY450139 orally once daily until Week 88.
  Interventions: Drug: LY450139
- 140 mg LY450139 (Experimental): Participants received 60 mg LY450139 orally once daily for 2 weeks, followed by 100 mg LY450139 orally once daily for 2 weeks, then 140 mg LY450139 orally once daily until Week 88.
  Interventions: Drug: LY450139

INTERVENTIONS:
Drug: LY450139 — Administered orally once daily
  Other Names: semagacestat
  Arms: 100 mg LY450139; 140 mg LY450139
Drug: Placebo — Administered orally once daily
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is a fatal degenerative disease of the brain for which there is no cure. AD causes brain cells to die. AD is thought to be caused by an excess of beta-amyloid (β-amyloid), a sticky protein in the brain that forms amyloid plaques. At autopsy, AD patients are required to have these amyloid plaques in the brain in order to have a definitive diagnosis of AD. Inhibiting the enzyme gamma-secretase (γ-secretase) lowers the production of β-amyloid. Semagacestat (LY450139) is a functional γ-secretase inhibitor and was shown to lower β-amyloid in blood and spinal fluid in humans tested thus far and in blood, spinal fluid, and brain in animals tested thus far. This study used several different tests to measure the effect of semagacestat on both β-amyloid and amyloid plaques for some participants. The build-up of amyloid plaques was measured by a brain scan that takes a picture of amyloid plaques in the brain. Other tests measured the overall function of the brain and brain size in some participants. In this trial, participants who initially received placebo (inactive sugar pill) were, at a certain point in the study, switched over to active drug, semagacestat. In other words, all participants could eventually receive active drug. Participation could last approximately 2 years. Participants taking approved AD medications were permitted to participate in this study and continue taking these medications during the study. All participants who completed this study had the option to continue receiving semagacestat by participating in an open-label study.

Preliminary results from this study (H6L-MC-LFAN [LFAN]) and another similar study (H6L-MC-LFBC [LFBC; NCT00762411]) showed semagacestat did not slow disease progression and was associated with worsening of clinical measures of cognition and the ability to perform activities of daily living. Study drug was stopped in all studies. Studies LFAN, LFBC, and open-label H6L-MC-LFBF (LFBF; NCT01035138) were amended to continue collecting safety data, including cognitive scores, for at least 7 months. The Clinical Trial Registry (CTR) will reflect results of analyses from the original LFAN protocol in addition to those from the amended LFAN protocol.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for mild to moderate Alzheimer's disease (AD) with Mini-Mental State Examination (MMSE) score of 16-26 at Visit 1
* Modified Hachinski Ischemia Scale score of less than or equal to 4
* Geriatric Depression Scale score of less than or equal to 6
* A magnetic resonance imaging (MRI) or computerized tomography (CT) scan in the last 2 years with no findings inconsistent with a diagnosis of AD
* If female, must be without menstruation for at least 12 consecutive months or have had both ovaries removed

Exclusion Criteria:

* Is not capable of swallowing whole oral medication
* Has serious or unstable illnesses
* Does not have a reliable caregiver
* Chronic alcohol or drug abuse within the past 5 years
* Has ever had active vaccination for AD

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1537 (Actual)
Dates: Start 2008-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours EST), Study Director — Eli Lilly and Company
Locations (147):
- United States (50):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sun City, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lomita, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamden, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooksville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pompano Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sunrise, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa Bay, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Yarmouth, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jenkintown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Providence, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bennington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Fe
- Australia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hornsby, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kogarah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Randwick, Sydney, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Geelong, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg West, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kew, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalst
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antwerp
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bruges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Penticton, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Chile (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antofagasta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concepción
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valdivia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viña del Mar
- Denmark (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roskilde
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Svendborg
- Finland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuopio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mikkeli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rouen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Regensburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siegen
- India (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kolkata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thiruvananthapuram
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tirupati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varanasi
- Israel (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashkelon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beersheba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Japan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukui
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokushima
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- South Africa (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellair
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., George
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johannesburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosebank
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Umhlanga
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albacete
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barakaldo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plasencia
- Sweden (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mölndal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norrköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uddevalla
- United Kingdom (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bath, Banes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southampton, Hants
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liverpool, Merseyside
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Swindon, Wilts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belfast
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newcastle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stoke-on-Trent

REFERENCES:
- [Derived] Liu-Seifert H, Siemers E, Price K, Han B, Selzler KJ, Henley D, Sundell K, Aisen P, Cummings J, Raskin J, Mohs R; Alzheimer's Disease Neuroimaging Initiative. Cognitive Impairment Precedes and Predicts Functional Impairment in Mild Alzheimer's Disease. J Alzheimers Dis. 2015;47(1):205-14. doi: 10.3233/JAD-142508. PMID 26402769
- [Derived] Henley DB, Dowsett SA, Chen YF, Liu-Seifert H, Grill JD, Doody RS, Aisen P, Raman R, Miller DS, Hake AM, Cummings J. Alzheimer's disease progression by geographical region in a clinical trial setting. Alzheimers Res Ther. 2015 Jun 25;7(1):43. doi: 10.1186/s13195-015-0127-0. eCollection 2015. PMID 26120369
- [Derived] Doody RS, Raman R, Sperling RA, Seimers E, Sethuraman G, Mohs R, Farlow M, Iwatsubo T, Vellas B, Sun X, Ernstrom K, Thomas RG, Aisen PS; Alzheimer's Disease Cooperative Study. Peripheral and central effects of gamma-secretase inhibition by semagacestat in Alzheimer's disease. Alzheimers Res Ther. 2015 Jun 10;7(1):36. doi: 10.1186/s13195-015-0121-6. eCollection 2015. PMID 26064192
- [Derived] Doody RS, Raman R, Farlow M, Iwatsubo T, Vellas B, Joffe S, Kieburtz K, He F, Sun X, Thomas RG, Aisen PS; Alzheimer's Disease Cooperative Study Steering Committee; Siemers E, Sethuraman G, Mohs R; Semagacestat Study Group. A phase 3 trial of semagacestat for treatment of Alzheimer's disease. N Engl J Med. 2013 Jul 25;369(4):341-50. doi: 10.1056/NEJMoa1210951. PMID 23883379
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo orally once daily for the first 76 weeks. At the end of 76 weeks, placebo arm participants received LY450139 titrated up to 140 mg orally once daily until Week 88.
Period: Initial Treatment
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Started | 501 | 507 | 529
Intent-to-treat (ITT) | 501 (ITT population included all randomized participants (pts) who had at least 1 dose of study drug.) | 506 (ITT population included all randomized participants who had at least 1 dose of study drug.) | 527 (ITT population included all randomized participants who had at least 1 dose of study drug.)
Completed | 189 | 153 | 121
Not Completed | 312 | 354 | 408
Not completed — Adverse Event | 51 | 121 | 144
Not completed — Death | 6 | 11 | 15
Not completed — Lost to Follow-up | 4 | 1 | 4
Not completed — Physician Decision | 3 | 2 | 4
Not completed — Protocol Violation | 2 | 2 | 5
Not completed — Withdrawal by Subject | 25 | 31 | 46
Not completed — Sponsor decision | 193 | 142 | 147
Not completed — Caregiver decision | 21 | 36 | 36
Not completed — Abnormal lab/electrocardiogram (ECG) | 7 | 7 | 6
Not completed — Entry criteria exclusion | 0 | 1 | 1
Period: Delayed Start
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Started | 189 | 153 | 121
Completed | 91 | 76 | 55
Not Completed | 98 | 77 | 66
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 12 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Caregiver Decision | 5 | 6 | 2
Not completed — Sponsor Decision | 77 | 66 | 59
Period: Safety Follow Up (SFU)-Optional
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Started | 290 (SFU was optional; pts entered from initial treatment and delayed start or did not enter SFU.) | 223 (SFU was optional; pts entered from initial treatment and delayed start or did not enter SFU.) | 214 (SFU was optional, pts entered from initial treatment and delayed start or did not enter SFU.)
Completed | 229 | 168 | 172
Not Completed | 61 | 55 | 42
Not completed — Death | 0 | 1 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 15 | 13
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Caregiver Decision | 17 | 16 | 9
Not completed — No safety visit or follow up | 25 | 22 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139 | Total
Number analyzed (Participants) | 501 | 506 | 527 | 1534
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (8.1) | 73.6 (8.0) | 73.9 (8.5) | 73.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278 | 279 | 263 | 820
  Male | 223 | 227 | 264 | 714
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 413 | 428 | 441 | 1282
  African | 3 | 6 | 3 | 12
  Hispanic | 33 | 22 | 24 | 79
  Native American | 0 | 0 | 2 | 2
  East Asian | 47 | 45 | 51 | 143
  West Asian | 5 | 5 | 6 | 16
Region of Enrollment [Number; unit: participants]
  United States | 192 | 194 | 199 | 585
  Finland | 6 | 8 | 8 | 22
  Spain | 24 | 24 | 25 | 73
  Chile | 17 | 14 | 12 | 43
  Israel | 22 | 21 | 21 | 64
  Italy | 6 | 5 | 6 | 17
  United Kingdom | 14 | 20 | 21 | 55
  India | 10 | 9 | 11 | 30
  France | 15 | 14 | 14 | 43
  Canada | 20 | 21 | 18 | 59
  Argentina | 24 | 23 | 26 | 73
  Poland | 12 | 15 | 18 | 45
  Belgium | 8 | 5 | 5 | 18
  Australia | 20 | 25 | 24 | 69
  Denmark | 5 | 5 | 4 | 14
  South Africa | 26 | 28 | 30 | 84
  Germany | 29 | 21 | 27 | 77
  Japan | 41 | 37 | 43 | 121
  Sweden | 10 | 17 | 15 | 42
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog11) Score [Mean (Standard Deviation); unit: units on a scale] — ADAS-Cog11 consists of 11 items assessing areas of function most typically impaired in AD: orientation, verbal memory, language, and praxis. The scale ranges from 0 to 70, with higher scores indicating greater disease severity.
  units on a scale | 22.8 (9.1) | 22.5 (8.9) | 23.1 (8.8) | 22.8 (8.9)
Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Inventory Score [Mean (Standard Deviation); unit: units on a scale] — The ADCS-ADL Inventory Score is a 23-item inventory developed as a Rater-administered questionnaire answered by the participant's caregiver. It measures performance of basic and instrumental activities of daily living by participants. The total ADCS-ADL score ranges from 0 to 78, with lower scores indicating greater disease severity.
  units on a scale | 60.5 (13.0) | 62.3 (11.6) | 60.5 (12.4) | 61.1 (12.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog11) Score at 76 Weeks
Description: ADAS-Cog11 was used as a primary efficacy measure. It consists of 11 items assessing areas of function most typically impaired in Alzheimer's disease (AD): orientation, verbal memory, language, and praxis. The scale ranges from 0 to 70, with higher scores indicating greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: The analysis population included all randomized participants who received at least 1 dose of study medication with baseline and at least 1 post baseline evaluable data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 270 | 216 | 199
units on a scale | 6.19 (0.54) | 7.29 (0.57) | 7.68 (0.59)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.134, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.610, Mixed Models Analysis

2. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog11) Score at 16 Weeks After Cessation of Study Drug
Description: ADAS-Cog11 consists of 11 items assessing areas of function most typically impaired in Alzheimer's disease (AD): orientation, verbal memory, language, and praxis. The scale ranges from 0 to 70, with higher scores indicating greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 16 weeks following treatment cessation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 204 | 154 | 146
units on a scale | 6.59 (0.80) | 7.57 (0.91) | 7.90 (0.90)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.296, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.172, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.746, Mixed Models Analysis

3. Primary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Inventory Score at 76 Weeks
Description: ADCS-ADL is a 23-item inventory developed as a Rater-administered questionnaire answered by the participant's caregiver. It measures performance of basic and instrumental activities of daily living by participants. The total score ranges from 0 to 78, with lower scores indicating greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 266 | 216 | 197
units on a scale | -8.76 (0.72) | -10.13 (0.77) | -12.70 (0.79)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.166, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis

4. Primary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Inventory Score at 16 Weeks After Cessation of Study Drug
Description: as for outcome 3
Time Frame: Baseline (randomization), 16 weeks following treatment cessation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 198 | 153 | 147
units on a scale | -9.26 (1.14) | -9.15 (1.28) | -11.73 (1.26)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.935, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.068, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.070, Mixed Models Analysis

5. Secondary Outcome: Percent Change From Baseline in Amyloid Beta (Aβ) 1-42 Plasma Concentration at 52 Weeks
Description: Concentration of amino acid peptide, known as Aβ 1-42, in plasma. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 309 | 265 | 245
picogram per milliliter (pg/mL) | 3.86 (2.32) | -5.97 (2.50) | -19.95 (2.58)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.002, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Secondary Outcome: Change From Baseline in Positron Emission Tomography (PET) Using Fluorine-18 Fluorodeoxyglucose (18F-FDG) at 76 Weeks
Description: Measurement of local cerebral glucose metabolism by PET using the radioactive tracer 18F-FDG. The outcome reported is the composite summary of the standard uptake value ratio (SUVR) normalized to the Pons. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 40 | 42 | 43
ratio | -0.08 (0.01) | -0.12 (0.01) | -0.11 (0.02)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.038, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.147, ANCOVA
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.604, ANCOVA

7. Secondary Outcome: Change From Baseline in Hippocampal Volume Using Volumetric Magnetic Resonance Imaging (vMRI) up to 76 Weeks
Description: The vMRI assessment of left and right hippocampal volume is reported. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cubic millimeter (mm^3)
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 75 | 69 | 64
cubic millimeter (mm^3)
  Left Hippocampal Volume | -96.54 (10.73) | -75.34 (11.06) | -107.62 (11.38)
  Right Hippocampal Volume | -108.69 (11.56) | -93.89 (12.19) | -112.40 (12.52)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.143, ANCOVA — This is the p-value for the Left Hippocampal Volume
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.464, ANCOVA — This is the p-value for the Left Hippocampal Volume
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.025, ANCOVA — This is the p-value for the Left Hippocampal Volume
Statistical Analysis 4: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.347, ANCOVA — This is the p-value for the Right Hippocampal Volume
Statistical Analysis 5: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.820, ANCOVA — This is the p-value for the Right Hippocampal Volume
Statistical Analysis 6: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.243, ANCOVA — This is the p-value for the Right Hippocampal Volume

8. Secondary Outcome: Change From Baseline in Amyloid Imaging Positron Emission Tomography (AV-45 PET) up to 76 Weeks
Description: A radioactive tracer for PET that is a ligand for amyloid called AV-45. This permits the visualization of amyloid in the brains of Alzheimer's participants. The outcome reported is the composite summary of the standard uptake value ratio (SUVR) normalized to the cerebellar gray matter. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 18 | 23 | 18
ratio | 0.08 (0.06) | 0.06 (0.06) | 0.09 (0.07)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.784, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.931, ANCOVA
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.718, ANCOVA

9. Secondary Outcome: Change From Baseline in Tau Concentration in Spinal Fluid up to 76 Weeks
Description: Concentration of total tau in spinal fluid. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 10 | 17 | 18
picogram per milliliter (pg/mL) | 75.11 (92.02) | 20.50 (69.54) | 61.00 (59.07)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.634, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.901, ANCOVA
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.659, ANCOVA

10. Secondary Outcome: LY450139 Population Pharmacokinetics: Clearance of LY450139
Description: Model estimated apparent oral clearance. Clearance is defined as the volume of plasma that is completely cleared of drug (LY450139) per unit time.
Time Frame: 6 weeks, 12 weeks, and 52 weeks
Population: The analysis population (N=974) included all participants randomized to LY450139 with sufficient drug concentration and dosing information to allow estimation of clearance.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Groups:
- LY450139: Participants received 60 mg LY450139 orally once daily for 2 weeks, followed by 100 mg LY450139 orally once daily for 2 weeks, then 140 mg LY450139 orally once daily until Week 88.
Arm/Group | LY450139
Number analyzed (Participants) | 974
liter per hour (L/h) | 18.8 (26.8)

11. Secondary Outcome: LY450139 Population Pharmacokinetics: Volume of Distribution of LY450139
Description: Model-estimated apparent volume of distribution. Volume of distribution is a measure of the extent to which the drug distributes in the body.
Time Frame: 6 weeks, 12 weeks, and 52 weeks
Population: The analysis population (N=974) included all participants randomized to LY450139 with sufficient drug concentration and dosing information to allow estimation of volume of distribution.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Groups:
- LY450139: Participants received 60 milligram LY450139 orally once daily for 2 weeks, followed by 100 mg LY450139 orally once daily for 2 weeks, then 140 mg LY450139 orally once daily until Week 88.
Arm/Group | LY450139
Number analyzed (Participants) | 974
liter (L) | 66.8 (26.1)

12. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog12) Score at 76 Weeks
Description: ADAS-Cog12 is ADAS-Cog11 augmented with delayed free recall measure, resulting in a total score ranging from 0 to 80. Higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 269 | 215 | 199
units on a scale | 6.52 (0.58) | 7.98 (0.61) | 8.33 (0.63)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.062, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.669, Mixed Models Analysis

13. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog14) Score at 76 Weeks
Description: ADAS-Cog14 is ADAS-Cog11 augmented with delayed free recall, digit cancellation, and maze completion measures. A score of 0 to 10 for delayed free recall and a conversion code of 0 to 5 for digit cancellation and maze completion provide total score ranges for this extended ADAS-Cog14 of 0 to 90. Higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 270 | 216 | 198
units on a scale | 7.42 (0.63) | 8.97 (0.67) | 9.48 (0.69)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.071, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.571, Mixed Models Analysis

14. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Score at 76 Weeks
Description: MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, and ability to name objects, follow verbal and written commands, write a sentence, and copy figures) in elderly participants. The total score ranges from 0 to 30; Lower score indicates greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 376 | 289 | 274
units on a scale | -2.95 (0.26) | -3.14 (0.27) | -3.71 (0.27)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.518, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.072, Mixed Models Analysis

15. Secondary Outcome: Change From Baseline in Clinical Dementia Rating-Sum of Boxes (CDR-SB) Score at 76 Weeks
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 267 | 216 | 195
units on a scale | 2.31 (0.17) | 2.73 (0.18) | 3.04 (0.18)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.069, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.198, Mixed Models Analysis

16. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Score at 76 Weeks
Description: NPI assesses psychopathology in participants with dementia and other neurologic disorders. Information is obtained from a caregiver familiar with the participant's behavior. Total score ranges from 12 to 144; Higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 369 | 298 | 271
units on a scale | 1.92 (0.75) | 3.31 (0.79) | 4.15 (0.81)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.127, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.381, Mixed Models Analysis

17. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional Health-Related Quality of Life Scale Proxy Version (EQ-5D Proxy) Visual Analog Scale (VAS) Score at 76 Weeks
Description: EQ-5D (proxy version) measures mobility, self-care, usual activities, pain/discomfort, anxiety/depression; each has 3 severity levels (no, some, severe problems) coded to a 1-digit number (1-3). Digits are combined into 5-digit number describing health state. Numerals 1-3 are not added for total score. VAS assesses caregiver's impression of participant's overall health state; scores range from 0 to 100; Lower scores indicate greater disease severity. Least Squares (LS) Mean value controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 374 | 300 | 275
units on a scale | -1.41 (1.11) | -7.49 (1.20) | -5.33 (1.22)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.141, Mixed Models Analysis

18. Secondary Outcome: Change From Baseline in Resource Utilization in Dementia-Lite (RUD-Lite) Score (Number of Hospitalizations) up to 76 Weeks
Description: Assesses healthcare resource utilization (formal and informal care). Information gathered on both caregivers (caregiving time, work status) and participants (accommodation and healthcare resource utilization) was collected from baseline and follow-up interviews; Reported number of hospitalizations per participant up to 76 weeks. Least Squares (LS) Mean value was controlled for age and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hospitalizations/participant
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 82 | 98 | 94
hospitalizations/participant | 0.55 (0.09) | 0.66 (0.07) | 0.83 (0.08)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.337, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.018, ANCOVA
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.157, ANCOVA

19. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog12) Score at 16 Weeks After Cessation of Study Drug
Description: as for outcome 12
Time Frame: Baseline (randomization), 16 weeks following treatment cessation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 204 | 154 | 146
units on a scale | 6.97 (0.84) | 8.27 (0.95) | 8.41 (0.94)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.186, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.149, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.889, Mixed Models Analysis

20. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog14) Score at 16 Weeks After Cessation of Study Drug
Description: as for outcome 13
Time Frame: Baseline (randomization), 16 weeks following treatment cessation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 204 | 153 | 146
units on a scale | 7.90 (0.93) | 9.30 (1.06) | 9.89 (1.04)
Statistical Analysis 1: Comparison: Placebo vs 100 mg LY450139; Test type: Superiority or Other; p = 0.202, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 140 mg LY450139; Test type: Superiority or Other; p = 0.075, Mixed Models Analysis
Statistical Analysis 3: Comparison: 100 mg LY450139 vs 140 mg LY450139; Test type: Superiority or Other; p = 0.616, Mixed Models Analysis

21. Secondary Outcome: Change From Baseline in Clinical Dementia Rating-Sum of Boxes (CDR-SB) Score at 4 Weeks After Cessation of Study Drug
Description: Semi-structured interview; Participant's cognitive status rated across 6 domains of functioning: memory, orientation, judgment/problem solving, community affairs, home/hobbies, personal care. Severity score assigned for each of 6 domains. Total score (SB) ranges: 0 to 18; Higher scores=greater disease severity. LS Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication. LY450139 dosing stopped due to evidence of dose-dependent cognitive/functional worsening. Participants followed off-dose for 32 weeks, but CDR-SB not assessed.
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: August 2010: all dosing was stopped after protocol-specified interim review showed dose-dependent cognitive/functional worsening of LY450139-treated participants. Participants were followed off-dose for 32 weeks. No analysis was performed at 4 weeks after cessation of drug since this outcome measure was not assessed during the follow-up period.
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Score at 4 Weeks After Cessation of Study Drug
Description: NPI assesses psychopathology in participants with dementia and other neurologic disorders. Information is obtained from a caregiver familiar with participant's behavior. Total score ranges from 12 to 144; Higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication. All LY450139 dosing stopped due to evidence of dose-dependent cognitive/functional worsening. Participants were followed off-dose for 32 weeks, but NPI was not assessed
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: as for outcome 21
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Score at 4 Weeks After Cessation of Study Drug
Description: MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, copy figures) in elderly participants. Total score ranges from 0 to 30; Lower score indicates greater disease severity. LS Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication. All LY450139 dosing was stopped due to evidence of dose-dependent cognitive/functional worsening. Participants were followed off-dose for 32 weeks, but MMSE was not assessed.
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: as for outcome 21
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional Health-Related Quality of Life Scale Proxy Version (EQ-5D Proxy) Visual Analog Scale (VAS) Score at 4 Weeks After Cessation of Study Drug
Description: EQ-5D (proxy version) measures mobility, self-care, usual activities, pain/discomfort, anxiety/depression. 3 severity levels: no, some, severe problems. VAS assesses caregiver's impression of participant's health state; score ranges from 0 to 100; Lower score indicates greater disease severity. LS Mean value controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication. All LY450139 dosing was stopped due to evidence of dose-dependent cognitive/functional worsening. Participants were followed off-dose for 32 weeks, but EQ-5D VAS was not assessed.
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: as for outcome 21
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Change From Baseline in Resource Utilization in Dementia-Lite (RUD-Lite) Score (Number of Hospitalizations) at 4 Weeks After Cessation of Study Drug
Description: RUD-Lite assesses healthcare resource utilization (formal and informal care). Information gathered on both caregivers (care-giving time, work status) and participants (accommodation, healthcare resource utilization) is collected. Reported number of participant hospitalizations. Least Squares (LS) Mean value controlled for age and investigator. All LY450139 dosing was stopped due to evidence of dose-dependent cognitive/functional worsening. Participants were followed off-dose for 32 weeks, but RUD-Lite was not assessed.
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: as for outcome 21
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Change From Baseline in Amyloid Beta (Aβ) 1-42 Concentration in Spinal Fluid up to 76 Weeks
Description: Concentration of an amino peptide known as Aβ 1-42 in spinal fluid. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 10 | 19 | 18
picogram per milliliter (pg/mL) | -86.16 (50.89) | 23.27 (34.55) | -40.51 (31.68)

27. Secondary Outcome: Change From Baseline in Phosphorylated-Tau (P-Tau) Concentration in Spinal Fluid
Description: Concentration of p-tau in spinal fluid. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | 100 mg LY450139 | 140 mg LY450139
Number analyzed (Participants) | 10 | 19 | 18
picogram per milliliter (pg/mL) | 9.75 (7.67) | -6.26 (5.46) | -5.13 (5.04)

ADVERSE EVENTS:
Description: Per statistical analysis plan, participants that had any visit for delayed start period were included in reporting of adverse events. Participants were not included in Participant Flow (PF), if they did not receive a dose during the delayed start period. Therefore, PF in delayed start period has less participant numbers than in Adverse Events.
Groups:
- Placebo - Initial Treatment Period (NT): Participants received placebo orally once daily for the first 76 weeks. At the end of 76 weeks, placebo arm participants received LY450139 titrated up to 140 milligrams (mg) orally once daily until Week 88.
- 100 mg LY450139 - NT; 100 mg LY450139 - DO: Participants received 60 mg LY450139 orally once daily for 2 weeks followed by gradual escalation to 100 mg LY450139 orally once daily until Week 88.
- 140 mg LY450139 - NT; 140 mg LY450139 - DO: Participants received 60 mg LY450139 orally once daily for 2 weeks, followed by 100 mg LY450139 orally once daily for 2 weeks, then 140 mg LY450139 orally once daily until Week 88.
- Placebo - Delayed Start Period (DO): Participants received placebo orally once daily for the first 76 weeks. At the end of 76 weeks, placebo arm participants received LY450139 titrated up to 140 mg orally once daily until Week 88.
- Placebo- Safety FU Period (SFU): For SFU, study drug had been stopped and period was optional to enter; Participants entered from Placebo initial treatment or delayed start or did not enter SFU.
- 100 mg LY450139- SFU: For SFU, study drug had been stopped and period was optional to enter; Participants entered from 100 mg LY450139 initial treatment or delayed start or did not enter SFU.
- 140 mg LY450139- SFU: For SFU, study drug had been stopped and period was optional to enter; Participants entered from 140 mg LY450139 initial treatment or delayed start or did not enter SFU.
Arm/Group | Placebo - Initial Treatment Period (NT) | 100 mg LY450139 - NT | 140 mg LY450139 - NT | Placebo - Delayed Start Period (DO) | 100 mg LY450139 - DO | 140 mg LY450139 - DO | Placebo- Safety FU Period (SFU) | 100 mg LY450139- SFU | 140 mg LY450139- SFU
Serious Adverse Events (participants affected / at risk) | 72/501 | 123/507 | 132/529 | 10/192 | 9/153 | 5/124 | 12/290 | 22/223 | 5/214
Other Adverse Events (participants affected / at risk) | 262/501 | 310/507 | 385/529 | 0/192 | 0/153 | 0/124 | 0/290 | 0/223 | 0/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Initial Treatment Period (NT) (N=501) | 100 mg LY450139 - NT (N=507) | 140 mg LY450139 - NT (N=529) | Placebo - Delayed Start Period (DO) (N=192) | 100 mg LY450139 - DO (N=153) | 140 mg LY450139 - DO (N=124) | Placebo- Safety FU Period (SFU) (N=290) | 100 mg LY450139- SFU (N=223) | 140 mg LY450139- SFU (N=214)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuropericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 14 (14) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyometra (Infections and infestations) | 0/278 (0) | 0/280 (0) | 1/263 (1) | 0/114 (0) | 0/85 (0) | 0/61 (0) | 0/168 (0) | 0/124 (0) | 0/107 (0)
Renal cyst infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Starvation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung squamous cell carcinoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/278 (0) | 1/280 (1) | 0/263 (0) | 0/114 (0) | 0/85 (0) | 0/61 (0) | 0/168 (0) | 0/124 (0) | 0/107 (0)
Pancreatic carcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/223 (0) | 0/227 (0) | 1/266 (1) | 0/78 (0) | 0/68 (0) | 0/63 (0) | 0/122 (0) | 1/99 (1) | 0/107 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/223 (1) | 0/227 (0) | 1/266 (1) | 0/78 (0) | 0/68 (0) | 0/63 (0) | 0/122 (0) | 0/99 (0) | 0/107 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/278 (0) | 0/280 (0) | 0/263 (0) | 1/114 (1) | 0/85 (0) | 0/61 (0) | 0/168 (0) | 0/124 (0) | 0/107 (0)
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/278 (0) | 1/280 (1) | 0/263 (0) | 0/114 (0) | 0/85 (0) | 0/61 (0) | 0/168 (0) | 0/124 (0) | 0/107 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain stem stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 7 (7) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delusional disorder, unspecified type (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis glandularis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral caruncle (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/223 (0) | 2/227 (2) | 1/266 (1) | 0/78 (0) | 1/68 (1) | 0/63 (0) | 0/122 (0) | 0/99 (0) | 0/107 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0/223 (0) | 0/227 (0) | 1/266 (1) | 0/78 (0) | 0/68 (0) | 0/63 (0) | 0/122 (0) | 0/99 (0) | 0/107 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immobile (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Initial Treatment Period (NT) (N=501) | 100 mg LY450139 - NT (N=507) | 140 mg LY450139 - NT (N=529) | Placebo - Delayed Start Period (DO) (N=192) | 100 mg LY450139 - DO (N=153) | 140 mg LY450139 - DO (N=124) | Placebo- Safety FU Period (SFU) (N=290) | 100 mg LY450139- SFU (N=223) | 140 mg LY450139- SFU (N=214)
Diarrhoea (Gastrointestinal disorders) | 54 (93) | 54 (67) | 71 (87) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 23 (27) | 51 (69) | 63 (71) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (21) | 44 (50) | 44 (67) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 30 (32) | 24 (25) | 31 (36) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 33 (40) | 24 (26) | 31 (33) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 19 (20) | 27 (33) | 31 (39) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 29 (39) | 31 (44) | 39 (44) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 40 (50) | 36 (45) | 33 (37) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 13 (14) | 25 (25) | 47 (48) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 16 (16) | 36 (37) | 56 (61) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 21 (21) | 32 (41) | 28 (30) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 35 (46) | 33 (42) | 41 (57) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 22 (23) | 27 (27) | 25 (27) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 15 (15) | 23 (23) | 35 (36) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 19 (21) | 26 (28) | 22 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 29 (36) | 35 (36) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 7 (8) | 63 (64) | 99 (106) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 9 (10) | 23 (25) | 28 (38) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 17 (20) | 36 (43) | 43 (50) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (8) | 16 (17) | 27 (28) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Outcomes with 4-week after study drug cessation timeframe=All dosing stopped after protocol-specified interim review showed dose-dependent cognitive/functional worsening for LY450139 participants; followed for 32 weeks; not all assessments were made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days